CLINICAL TRIAL: NCT05298943
Title: Relation Between Cortical Activation and Graded Force Level During Robot-assistance Walking in Healthy People : A Functional Near-infrared Spectroscopy Neuroimaging Study.
Brief Title: Exoskeleton and Brain Activity With fNIRS
Acronym: ExoNIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHRO-2021-11
Record Dates: First submitted 2022-03-16; First posted 2022-03-28 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Healthy; Gait Disorders, Neurologic
Keywords: fNIRS; Motor cortex activity; Gait; Effort; exoskeleton
MeSH Terms: conditions — Gait Disorders, Neurologic | interventions — Walking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with 4 walking situations (Other)
  Interventions: Other: walking in 4 situations

INTERVENTIONS:
Other: walking in 4 situations — Recording of cerebral hemodynamic with fNIRS during gait in exoskeleton with Four strength levels of aid : total aid (A100%), partial aid (A50%), no aid (A0%) and resistance of 25 % (R25%) to walking from the exoskeleton. Each subject are recorded during 8 trials for each level (32 trials). The order is counterbalanced among the subjects

SUMMARY:
Background. Force control is one of the major parameter of motor activity. There is few study concerning the cortical activity imply for different levels of force during gait.

Objective. To investigate cortex activation while walking an exoskeleton with 4 levels of guidance force in healthy controls.

Methods. The investigators acquired near-infrared spectroscopy (fNIRS) with a 20 channels device (Brite 24® ; Artinis) covering bilaterally most motor control brain regions during exoskeleton walking at different level of force (100 %, 50% aid, 0 % aid and 25 % of resistance) in 24 healthy controls. The investigators measured variations of oxyhemoglobin (HbO2) and deoxyhemoglobin (HbR). The technique was optimized by the use of reference channels (to correct for superficial hemodynamic interference).

DETAILED DESCRIPTION:
An important goal of motor systems neuroscience is to characterize how neural activity in the brain mediates movement parameters such as force, velocity, frequency of movement or movement direction. The neural codage of force has been studied in animal and human with TEP , fMRI , functional near-infrared spectroscopy (fNIRS), EEG or magnetic stimulation.

Electrophysiological studies in nonhuman primates demonstrated a correlation between neuronal discharge rates in multiple regions of the contralateral motor cortex and exerted force amplitude .

In humans, functional magnetic resonance imaging (fMRI) studies confirmed the relation between increasing neuronal activation and increasing amplitude of force in the contralateral primary motor/somatosensory (M1/S1) cortices, supplementary motor area (SMA), and premotor cortex. The ipsilateral motor cortex could also contribute to the force codage. There are also evidences that the basal ganglia-thalamo-cortical loop participates to the regulation of force control. The internal portion of the globus pallidus (GPi) and subthalamic nucleus (STN) had a positive increase in percent signal change with increasing force, and the ventral thalamic regions were also implied in the the same way. More recently, studies with fNIRS confirmed the relationship between force level and cerebral activation in contralateral and ipsilateral hemisphere.

Most of the human studies concerned isometric static tasks. Only few studies considered dynamic movements. As a rule, the processing of repetitive transient force changes requires more metabolic activity than the generation and control of a static force. There is a correlation between the force level and cortical changes within the neuronal network in contralateral M1 and anterior cerebellum.

Most of the studies concern the upper limb. To our knowledge only to studied concern the lower limb in an isometric force level. One concerns the neural correlates of quadriceps torque control in chronic obstructive pulmonary disease patients and the other one concerns isometric contractions with the ankle dorsiflexor in healthy controls.

fMRI and TEP are highly sensitive to motion artifacts and not suitable for dynamic proximal joints or gait studies. fNIRS is less sensitive to motion artifacts and has permitted numerous studies of walking under more natural conditions in controls or patients. fMRI and fNIRS are based on the physiological principles of neurovascular coupling, the process by which active brain regions induce a local increase in blood flow to match their energy demands via the dilation of capillaries and arterioles. fMRI measures the blood oxygen level-dependent (BOLD) response corresponding to the ratio of oxy to deoxy-hemoglobin. However, the two moieties of hemoglobin are not individually measured with fMRI. On the contrary, fNIRS measures the two hemoglobin species separately. During this neurovascular coupling, the amount of oxygen supplied is typically greater than that consumed locally, resulting in a substantial increase in HbO2 and a slight reduction in HbR in the region.

Many of the fNIRS studies about gait recorded hemodynamic variations in the prefrontal cortex with dual tasks paradigm. Only few studies concerned the motor cortex.

In recent years, robot-assisted rehabilitation has been used in addition to conventional rehabilitation. It offers opportunities for early, intensive, task-specific management with multi-sensory stimulation that is considered the most efficient for promoting neuroplasticity. Literature suggests that robotic rehabilitation increases the walking ability of patients , walking speed , lower limb muscle strength, step length and walking symmetry . However, the neurophysiological bases of robot-assisted rehabilitation remain poorly known. The use of an exoskeleton makes it possible to control the percentage of aid provided. In this study in healthy subjects the investigators propose to study brain activation in motor regions when walking in an exoskeleton. Four strength levels are studied: total aid (A100%), partial help (A50%), no help (A0%) and resistance of 25 % (R25%) to walking from the exoskeleton. The investigators hypothesize that the level of brain activation measured by fNIRS will increase with the effort provided by the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (with no known neurological, rheumatological or cardiological medical history)
* Age between 18 and 40
* Having social security coverage,
* Having given written consent.
* Height > 1.5 meters
* Weight less than 100 kg.
* Respect of the morphological criteria

Exclusion Criteria:

* Person under guardianship or curatorship,
* Walking with assistance,
* Trauma or orthopedic disorder that may affect walking,
* Pregnant women,
* Medication that alters alertness and potentially affects walking and attentional abilities,

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Change of oxyhemoglobin concentration during gait tasks | Day 0
Change of desoxyhemoglobin concentration during gait tasks | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AUZOU, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR Orléans, Boissise-le-Roi, France

REFERENCES:
- [Background] Chen WL, Wagner J, Heugel N, Sugar J, Lee YW, Conant L, Malloy M, Heffernan J, Quirk B, Zinos A, Beardsley SA, Prost R, Whelan HT. Functional Near-Infrared Spectroscopy and Its Clinical Application in the Field of Neuroscience: Advances and Future Directions. Front Neurosci. 2020 Jul 9;14:724. doi: 10.3389/fnins.2020.00724. eCollection 2020. PMID 32742257
- [Background] Kim H. Corrigendum to "Cerebral hemodynamics predicts the cortical area and coding scheme in the human brain for force generation by wrist muscles" [Behav. Brain Res. 396 (2021) 112865]. Behav Brain Res. 2021 Feb 26;400:113054. doi: 10.1016/j.bbr.2020.113054. Epub 2020 Dec 17. No abstract available. PMID 33341645